CLINICAL TRIAL: NCT00720005
Title: Evaluation of the Aspheric ReSTOR IOL After Routine Cataract Extraction
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Kerry D Solomon, MD, Storm Eye Institute - Medical University of South Carolina
Other Study IDs: MRC-07-002
Record Dates: First submitted 2008-07-18; First posted 2008-07-22 (Estimated); Last update posted 2010-10-04 (Estimated); Status verified 2010-10

CONDITIONS: Cataract
Keywords: Cataract; cataract extraction; intraocular lens; age related
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Aspheric Acrysof ResTOR Lens: Implantation of Aspheric Acrysof ResTOR
  Interventions: Device: Aspheric Acrysof ReSTOR intraocular lens

INTERVENTIONS:
Device: Aspheric Acrysof ReSTOR intraocular lens — Bilateral implantation of Aspheric Acrysof ReSTOR
  Other Names: Acrysof ReSTOR

SUMMARY:
The purpose of this study is to evaluate the visual outcomes and patient satisfaction after bilateral implantation of the aspheric ReSTOR multifocal intraocular lens (IOL) and compare it to a historical control group of patients implanted bilaterally with the spherical ReSTOR multifocal

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the visual outcomes and patient satisfaction after bilateral implantation of the aspheric ReSTOR multifocal intraocular lens (IOL) and compare it to a historical control group of patients implanted bilaterally with the spherical ReSTOR multifocal.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have an age-related cataract in both eyes.
* 40 years of age or older.
* Patient must desire cataract extraction.
* Expected maximum of 2 weeks and minimum of 1-week interval between first and second eye surgeries.
* Willing and able to comply with scheduled visits and other study procedures

Exclusion Criteria:

* Preoperative ocular pathology potentially affecting visual acuity.
* Keratometric astigmatism exceeding 1.50 diopters.
* Planned postoperative refraction for mono-vision.
* Uncontrolled diabetes.
* Use of any systemic or topical drug known to interfere with visual performance.
* Contact lens use during the active treatment portion of the trial.
* Any concurrent infectious/non infectious conjunctivitis, keratitis or uveitis.
* Pregnant or nursing mothers and females of childbearing potential not practicing a reliable and medically acceptable method of birth control.
* Any clinically significant, serious or severe medical or psychiatric condition that may increase the risk associated with study participation or study device implantation or may interfere with the interpretation of study results.
* Participation in (or current participation) any investigational drug or device trial within the previous 30 days prior to the start date of this trial.
* Intraocular conventional surgery within the past three months or intraocular laser surgery within one month in the operated eye.
* Other ocular surgery at the time of the cataract extraction.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects 18 years or older who had cataract surgery.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2007-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
ETDRS uncorrected and best corrected visual acuity at distance, intermediate, and near, manifest refraction, distance corrected near visual acuity (DCNVA), and best near point (optimal reading distance). | Preoperatively, 1, 3 and 6 months postoperatively

SECONDARY OUTCOMES:
pupil size and contrast sensitivity under photopic and mesopic conditions wearing the best distance correction (the latter per eye and both eyes. Slit-lamp exam, eye dominance, reading speed test, and a quality of vision questionnaire. | preoperatively, 1, 3, 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Kerry D. Solomon, MD, Principal Investigator — Assistant Professor
Locations (1):
- Storm Eye Institute, Medical University of South Carolina, Charleston, South Carolina, United States